CLINICAL TRIAL: NCT02414867
Title: Total Energy Expenditure and Fat Oxidation in 2 Year Old Children
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 203770
Record Dates: First submitted 2015-04-08; First posted 2015-04-13 (Estimated); Last update posted 2024-11-25 (Actual); Status verified 2023-12

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine collected
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Normal weight mothers
- 2: Overweight/Obese mothers

SUMMARY:
The purpose of the study is to determine energy expenditure and fat oxidation in 2 year old children.

ELIGIBILITY:
Inclusion Criteria:

* 1.5-2.5 years of age
* Mother is a participant of the Glowing study (NCT01131117)
* Healthy without taking medication that can affect study outcomes, as determined by the PI

Exclusion Criteria:

* None listed

Ages: 2 Years to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 120 toddlers born from mothers of the Glowing study (NCT01131117)
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2015-02; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
To determine total energy expenditure in 2 year old children | 15 days
  Doubly labeled water is administered to 2 year old children and urine is collected at different time points.
To determine fat oxidation in 2 year old children | 2-6 hours
  Deuterated palmitate is administered and urine is collected at different time points.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabet Borsheim, PhD, Principal Investigator — Arkansas Children's Nutrition Center
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States